CLINICAL TRIAL: NCT02046629
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetic Profiles of 14 mg Teriflunomide Tablet in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetic Profiles of Single 14 mg Teriflunomide Tablet in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PKM12788; U1111-1152-4217 (Other: UTN)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Cholestyramine Resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- teriflunomide dose 1 (Experimental): Teriflunomide 14mg tablet, oral single dose, fast condition Cholestyramine power, 8 gram,oral three times a day for 4 days, fed condition
  Interventions: Drug: Teriflunomide HMR1726; Drug: cholestyramine

INTERVENTIONS:
Drug: Teriflunomide HMR1726 — Pharmaceutical form:tablet Route of administration: oral
Drug: cholestyramine — Pharmaceutical form:power Route of administration: oral

SUMMARY:
Primary Objective:

To assess the pharmacokinetic (PK) parameters of teriflunomide after a single oral dose of 14 mg administration in Chinese healthy subjects

Secondary Objective:

To assess the safety and tolerability after a single oral dose of 14 mg teriflunomide in Chinese healthy subjects

DETAILED DESCRIPTION:
* Screening: 2 to 21 days before inclusion (Day -21 to Day -2)
* Institutionalization period: 6 days including 1 treatment day (Day -1 to Day 6, treatment on Day 1)
* Follow-up: 7-10 days (may be extended)
* End of study: Day 38 to Day 41 (may be extended)
* Total study duration: maximum 9 weeks

ELIGIBILITY:
Inclusion criteria :

Male or female subjects, between 18 and 45 years of age, inclusive. Body weight between 50.0 and 95.0 kg, inclusive, if male, and between 45.0 and 85.0 kg, inclusive, if female, body mass index between 19.0 and 24.0 kg/m2, inclusive.

Certified as healthy by a comprehensive clinical assessment and lab test. Subject must use an appropriate contraception method. Having given written informed consent prior to any procedure related to the study.

Exclusion criteria:

Blood donation, any volume, within 3 months before inclusion. Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined by a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from the supine to the standing position.

Excessive consumption of beverages with xanthine bases (>4 cups or glasses per day).

If female, pregnancy (defined as positive β-hCG blood test), breast-feeding. Any medication (including St John's Wort and traditional Chinese herb medicine) within 14 days before the inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of that drug, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days.

Any consumption of citrus (grapefruit, orange, etc) or their juices within 5 days before inclusion.

Subject (both male and female) who disagrees to use an appropriate contraception method .

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for teriflunomide determined from plasma concentration | 5 weeks

SECONDARY OUTCOMES:
safety assessments (adverse events, laboratory data, vital sign, and ECG parameters) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 156001, Shanghai, China